CLINICAL TRIAL: NCT00010309
Title: Phase I/II Trial Investigating The Safety And Immunogenicity Of Adenoviruses Encoding The Melan-A/MART-1 And gp 100 Melanoma Antigens Administered Intradermally To Patients With Stage II-IV Melanoma
Brief Title: Vaccine Therapy in Treating Patients Who Have Stage II, Stage III, or Stage IV Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068478; GENZ-ADVMEL-001-99; DFCI-00069; GENZ-2000-P-000380/1
Record Dates: First submitted 2001-02-02; First posted 2003-11-11 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-07

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen

INTERVENTIONS:
Biological: MART-1 antigen
Biological: gp100 antigen

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy in treating patients who have stage II, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and the maximum tolerated dose of vaccines containing two adenoviral vectors encoding the melanoma antigens Melan-A/MART-1 and gp100 in patients with stage II-IV melanoma. II. Assess the dose-response changes in the frequency of MART-1 and gp100 reactive T cells (CD4+ and CD8+) in patients receiving one of three different vaccine regimens. III. Assess the T-cell response to one melanoma antigen following three treatments with the other antigen in these patients. IV. Assess the effect of concomitant vaccination with both antigens on T-cell response in these patients.

OUTLINE: This is a dose escalation study. Patients are sequentially enrolled on 1 of 3 treatment arms. Each treatment arm has 3 groups. Arm I: Patients receive Ad2/MART-1v2 vaccine and Ad2/gp100v2 vaccine intradermally (ID) at the lowest dose level once every three weeks for either 6 or 15 weeks depending on assignment. Arm II: Patients receive Ad2/gp100v2 vaccine and Ad2/MART-1v2 vaccine ID at the mid-range dose level once every three weeks for either 6 or 15 weeks depending on assignment. Arm III: Patients receive Ad2/MART-1v2 vaccine and Ad2/gp100v2 vaccine ID at the highest dose level once every three weeks for either 6 or 15 weeks depending on assignment. Cohorts of 3-6 patients receive escalating doses of Ad2/MART-1v2 and/or Ad2/gp100v2 vaccines in each arm until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Patients are followed at 3 months, 6 months, and 1 year after completion of treatment.

PROJECTED ACCRUAL: A total of 24-36 patients will be accrued over 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage II, III, or IV cutaneous malignant melanoma No evidence of disease at time of entry to protocol Definitive complete surgical resection within past 12 months HLA-A2 positive

PATIENT CHARACTERISTICS: Age: 18 or over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,000 cells/mm3 Platelet count at least 100,000 cells/mm3 No clinically significant hematologic disease that would preclude study Hepatic: SGOT and SGPT less than 2 times upper limit of normal Bilirubin less than 2 mg/dL No clinically significant hepatic disease that would preclude study Renal: Creatinine less than 2 mg/dL No clinically significant renal disease that would preclude study Cardiovascular: No clinically significant cardiac disease that would preclude study Other: No clinically significant underlying condition that would preclude study No significant autoimmune disease or other major immune system disorder HIV negative HTLV negative Hepatitis B and C negative No active infection requiring parenteral antibiotics No psychiatric disorder that could hinder protocol compliance Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior or concurrent immunotherapy At least 3 months since prior interferon therapy Chemotherapy: No prior or concurrent chemotherapy Endocrine therapy: No prior or concurrent immunosuppressants Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 4 weeks since prior surgery Other: No other prior or concurrent experimental anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: Amy E. Bock, Study Chair — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Genzyme Corporation, Cambridge, Massachusetts
  - U.S. Oncology, Houston, Texas